CLINICAL TRIAL: NCT04060875
Title: Research Protocol for Karuna Labs Inc.: Safety and Efficacy of Virtual Reality Graded Motor Imagery for Chronic Pain
Status: Completed | Type: Observational
Sponsor: Karuna Labs Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAIRB-17-0063
Record Dates: First submitted 2019-07-29; First posted 2019-08-19 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pain; Low Back Pain; Fibromyalgia; Upper Extremity Dysfunction; Complex Regional Pain Syndromes; Phantom Limb Pain; Rheumatoid Arthritis; Carpal Tunnel Syndrome; Repetitive Strain Injury
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Fibromyalgia; Complex Regional Pain Syndromes; Phantom Limb; Arthritis, Rheumatoid; Carpal Tunnel Syndrome; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Feasibility group: First phase group will involve piloting a novel virtual reality treatment for chronic pain to investigate feasibility and safety with a smaller number of patients
  Interventions: Device: Karuna Labs Virtual Reality Software

INTERVENTIONS:
Device: Karuna Labs Virtual Reality Software — The subjects will engage in the three therapeutic modules: laterality, motor imagery, and 'mirroring.' The decision of which module to employ will be based on the subject's readiness and comfort on a case-by-case basis. A subject visit can be expected to last 40 minutes, with enough time to complete PHQ-9, and to accustom to the virtual reality setup by playing in a non-therapeutic virtual environment should they choose to do so. Time in the virtual reality is expected to last approximately 20 minutes per session.

SUMMARY:
The purpose of this study is to investigate, in two phases: (1) the feasibility and safety of Virtual Embodiment Therapy in treating chronic pain of lower back and upper limbs and (2) the efficacy of Virtual Embodiment Therapy on chronic pain disorders of the lower back and upper limbs. In phase 1, we will investigate the feasibility, safety, and side effects related to this treatment by assessing simulator sickness. In phase 2, which in contingent on successful completion of phase 1, we will assess symptoms of pain specific to the region treated, fear and avoidance behavior, and depression symptoms before and after 8 sessions of treatment with Virtual Embodiment Therapy in order to assess efficacy. This study will be single-blinded, because the participation of the clinician is necessary to ensure proper administration of the therapy, as well as to monitor in the event of adverse reactions.

DETAILED DESCRIPTION:
This multi-site study aims to investigate the feasibility, safety, and efficacy of using embodied virtual reality graded motor imagery software to treat adults with diagnosed chronic central pain conditions in two bodily regions: chronic pain in the lower back and in the upper limbs. The research will be conducted in two phases, the second of which is contingent upon successful completion of the first. The first phase will involve piloting a novel virtual reality treatment for chronic pain to investigate feasibility and safety with a smaller number of patients (N=30 for each condition). The second phase of the research will investigate efficacy using a single-blinded randomized control study design with sham control. Chronic pain conditions of the lower back and upper limbs will be investigated separately, and power analyses have been conducted to determine optimal study size, which is N=200 for each portion.

Central pain is defined as pain that originates in the central nervous system, and is not immediately due to injury, but is possibly a delayed reaction to injury. Example conditions eligible for this study include chronic lower back pain, as well as phantom limb pain, complex regional pain syndrome, carpal tunnel syndrome, post-stroke limb pain, and repetitive strain injuries of the shoulder, arm or hand. In the pilot phase of the study, 30 subjects with chronic lower back pain and 30 subjects with chronic upper limb pain will receive 8 sessions of graded motor imagery virtual reality therapy. Contingent on the success of the pilot, defined as completion of 8 session with no adverse events, and trends indicating improvement of range of motion, pain, fear/avoidance, and depression symptoms, the randomized control trial phase of the research will proceed. In the randomized phase, subjects will be randomized into active or control conditions. Active condition subjects will receive 8 sessions of graded motor imagery in virtual reality, and control condition subjects will receive a non-embodied sham virtual reality experience. This study will investigate the safety and feasibility of this approach, as well as its effects on pain symptoms.

This product is considered a non-significant risk device, as is explained in the accompanying letter from the sponsor, Karuna Labs Inc. A request for feedback from the presubmission program of the U.S. Food and Drug Administration has additionally been submitted.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the English language
2. Have had a chronic central pain of the lower back or upper limbs diagnosis for 3 months or longer
3. Can attend sessions at the study center twice a week for 4 weeks
4. Able to wear a VR HMD (head-mounted display) and move head in cervical rotation, extension, and flexion

Exclusion Criteria:

1. Individuals with a history of Severe Mental Illness, including schizophrenia, bipolar disorder I or II, or PTSD
2. History of susceptibility to seizures per subject's reporting
3. Pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People diagnosed with chronic pain disorders of the lower back or upper limbs with a continual duration of at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 1-2 months
  Safety and feasibility
Simulator Sickness Questionnaire | 1-2 months
  The questionnaire asks participants to score 16 symptoms on a four point scale (0-3). The scale measures susceptibility to nausea, general discomfort, stomach awareness, sweating, increased salivation, vertigo, burping, dizziness with eyes open, fullness of head, dizziness with eyes closed, difficulty focusing, headache, blurred vision, fatigue, and eye strain
Visual Analogue Scale (VAS) | 1-2 months
  The pain Visual Analogue Scale is a unidimensional measure of pain intensity. Patients are asked to rate the intensity of their pain using a horizontal line 10 centimeters (100 mm) in length. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])

SECONDARY OUTCOMES:
Fear and Avoidance Beliefs Questionnaire | 1-2 months
  The Fear and Avoidance Beliefs Questionnaire is a questionnaire based on the Fear-Avoidance Model of Exaggerated Pain Perception. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear-avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)
OSWESTRY Disability Index Questionnaire | 1-2months
  A patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those with low back pain. Questionnaire examines perceived level of disability in 10 everyday activities of daily living concerning the intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.
Pain Catastrophizing Scale | 1-2 months
  The Pain Catastrophizing Scale is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). The PCS is broken into three subscales being magnification, rumination, and helplessness. The scale was developed as a self-report measurement tool that provided a valid index of catastrophizing in clinical and non-clinical populations
Patient Health Questionnaire | 1-2 months
  The Patient Health Questionnaire is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 consists of 9 items of DSM-IV criteria as "0" (not at all) to "3" (nearly every day)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trujillo, PhD, Principal Investigator — Vice President of Clinical Affairs
Locations (1):
- Remedy Medical Group, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saby A, Alvarez A, Smolins D, Petros J, Nguyen L, Trujillo M, Aygun O. Effects of Embodiment in Virtual Reality for Treatment of Chronic Pain: Pilot Open-Label Study. JMIR Form Res. 2024 Feb 16;8:e34162. doi: 10.2196/34162. PMID 38363591